CLINICAL TRIAL: NCT00403091
Title: Internet Intervention to Improve Rural Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Carlos Estrada, UAB
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: X050111012; R18DK065001 (NIH)
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes mellitus; Internet; Education, Professional; Quality Indicators, Health Care; Quality of Health Care; Hypertension; Hyperlipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypertension; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Internet Intervention
- Control (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Internet Intervention — Internet-based intervention aims to improve guideline adherence by rural physicians caring for adult patients with type 2 diabetes.
  Arms: Intervention
Behavioral: Control — The comparison group will receive a text-based, non-interactive Internet posting of publicly available resources.
  Arms: Control

SUMMARY:
Rural Diabetes Online Care (RDOC) will develop an Internet-based intervention for rural primary care physicians, focusing on improving care for adult patients with diabetes. The intervention, drawing upon the principles of quality improvement and providing tools for system-based changes in practice, is designed for the rural practice, where resources are constrained.

DETAILED DESCRIPTION:
This 4-year randomized trial of an Internet-based intervention aims to improve guideline adherence by rural physicians caring for adult patients with type 2 diabetes.

Objectives. (1) Assess barriers to implementation of diabetes guidelines and identify solutions through focus groups and case-based vignette surveys; (2) Develop and implement an interactive Internet intervention including individualized physician performance feedback; (3) Evaluate the intervention in a randomized controlled trial; and (4) Examine the sustainability of improved guideline adherence once feedback ceases.

Methods. In partnership with the University of Alabama rural medicine program, we will randomize 200 rural physician offices to an intervention or comparison arm. Our 18-month intervention, customized to the individual physician in real-time, consists of Internet learning modules with case-based education, performance feedback, and benchmarks. The comparison group will receive a text-based, non-interactive Internet posting of publicly available resources. Nurse practitioners and physician assistants from the offices of study physicians may also participate in the Internet modules. Outcomes will be based on previously developed and validated quality measures for diabetes. The intervention will cover screening, diagnosis, treatment, and prevention. Performance feedback will include 10-15 charts per intervention physician. The main analysis, conducted at the physician level, will compare differential improvement in guideline adherence between the study arms. Ancillary analyses will examine the effects of physician characteristics, other providers in the office, and patient characteristics (e.g., comorbidities, ethnicity, gender, age, and socioeconomic status). Multivariable techniques will adjust for repeated measures, clustering of patients within physicians, and multiple providers within a single office.

Study Population. RDOC will enroll 200 physicians from rural Alabama, Mississippi, Georgia, Tennessee, Florida, Arkansas, Kentucky, North Carolina, South Carolina, Missouri, and West Virginia. Participating physicians will be randomized to receive the intervention or to a comparison group, which will receive traditional, text-based continuing medical education (CME). Each participating physician will allow two rounds of medical record abstraction to be conducted in his/her office. Results from the medical record review: (1) be used in the intervention to provide physicians with personal performance feedback and (2) used to examine change in performance for the intervention and comparison physicians as an evaluation of the entire study.

Significance. This study offers a technologically advanced, theory-grounded intervention for improving care of a high-risk, underserved population. With expertise in translating research into practice, rural medicine, behavioral medicine, health informatics, and clinical diabetes, our multidisciplinary team has a proven record of collaboration. This project will produce an evidence-based and replicable intervention that can be sustained in the "real world," and easily modified for other diseases. This project is substantially improved after making important changes recommended in the second review.

ELIGIBILITY:
Inclusion Criteria:

* Rural Primary Care Physicians

Exclusion Criteria:

* Non-rural non-primary care physicians

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2005-04; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
A1c | January 2005-present
Blood Pressure | January 2005-present
Lipids | January 2005-present

SECONDARY OUTCOMES:
Eye screening | January 2005-present
Foot exam | January 2005-present
Kidney disease monitored | January 2005-present
Dietary or exercise advice | January 2005-present
Smoking cessation advice | January 2005-present

CONTACTS AND LOCATIONS:
Overall Officials: Jeroan J Allison, MD, MS Epi, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama, Tuscaloosa, Alabama

REFERENCES:
- [Background] Safford MM, Allison JJ, Kiefe CI. Patient complexity: more than comorbidity. the vector model of complexity. J Gen Intern Med. 2007 Dec;22 Suppl 3(Suppl 3):382-90. doi: 10.1007/s11606-007-0307-0. PMID 18026806
- [Result] Safford MM, Shewchuk R, Qu H, Williams JH, Estrada CA, Ovalle F, Allison JJ. Reasons for not intensifying medications: differentiating "clinical inertia" from appropriate care. J Gen Intern Med. 2007 Dec;22(12):1648-55. doi: 10.1007/s11606-007-0433-8. Epub 2007 Oct 24. PMID 17957346
- [Result] Foster PP, Williams JH, Estrada CA, Higginbotham JC, Voltz ML, Safford MM, Allison J. Recruitment of rural physicians in a diabetes internet intervention study: overcoming challenges and barriers. J Natl Med Assoc. 2010 Feb;102(2):101-7. doi: 10.1016/s0027-9684(15)30497-1. PMID 20191922
- [Derived] Billue KL, Safford MM, Salanitro AH, Houston TK, Curry W, Kim Y, Allison JJ, Estrada CA. Medication intensification in diabetes in rural primary care: a cluster-randomised effectiveness trial. BMJ Open. 2012 Sep 17;2(5):e000959. doi: 10.1136/bmjopen-2012-000959. Print 2012. PMID 22991217
- See also: Rural Diabetes Online Care Project Website — http://www.ruraldoc.org